CLINICAL TRIAL: NCT03737487
Title: Effectiveness of the Montpellier Falls Clinic in Preventing Injuries in Older High-risk Adults
Brief Title: Effectiveness of the Montpellier Falls Clinic in Preventing InjuRiEs
Acronym: EMPIRE
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0393
Record Dates: First submitted 2018-11-02; First posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Falls
Keywords: geriatric assessment; fear of falling; injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Multidisciplinary fall risk and geriatric comprehensive assessment — * Complete blood count, serum electrolytes, C-Reactive Protein, transaminases and gamma-glutamyl transferase, thyroid-stimulating hormone, and 25OH vitamin D.
  * Calculation of BMI
  * A 40-min assessment of balance, walking speed, muscle strength, activity, and functional status by a physiotherapist
  * A 40-min assessment by an occupational therapist, including a detailed questionnaire on social support, living situation and home environment, fear of falling, and cognitive function
  * A 20-min assessment by a podiatrist including an examination of the patient's feet and footwear.
  * A 60-min assessment by a geriatrician including assessment of circumstances of the previous fall(s), review of current medications and medical history, and an in-depth examination of the patient to detect possible contributors or risk factors for falling
  * A 20-min review meeting with the 4 healthcare professionals in order to prioritize recommendations to be provided.

SUMMARY:
A falls prevention clinic opened in Montpellier (France) in 2015. The objective of the project is to evaluate whether the tailored multifactorial programme delivered in this real practice setting by a geriatrician, a podiatrist, a physiotherapist, and a occupational therapist would help prevent injuries in high-risk older patients using a 6-month pre-post intervention analysis.

DETAILED DESCRIPTION:
The Montpellier falls prevention clinic is a referral-based clinic specialized in the prevention of falls and fractures among patients aged 65+ (http://www.chu-montpellier.fr/fr/crepc/). The FPC that opened in 2015 is a member of the European Commission in its European Innovation Partnership on Active and Healthy Ageing (EIP on AHA) A2 action plan. The main mission of the clinic is to identify the underlying causes of the patients' falls, and to address modifiable risk factors in collaboration with family physicians in order to prevent injurious falls.

Based on a geriatric assessment performed by a geriatrician, a podologist, a occupational therapist, and a physiotherapist, the likely diagnoses and recommendations are notified in the medical report that is handed over to the patient or the caregiver for the patient's GP, along with the prescriptions, and sent also by mail to the GP. Recommendations remain under the GP's control with the possibility of another consultation if needed.

All patients admitted to the FPC are reassessed by phone at 3 months to register falls and injuries, and at 6 months to register falls and injuries, assess fear of falling, mobility and ability to perform activities of daily living, and satisfaction for the programme, and list proposed measures effectively applied.

ELIGIBILITY:
Inclusion Criteria:

All patients aged 65 or older with a history in the previous year of recurrent falls, or of a fall associated with a balance, gait, or muscle strength problem referred to the Montpellier falls prevention clinic

Exclusion Criteria:

* patients unable to walk 3 metres with or without an assistive device
* patients expected to live for less than 6 months based on the geriatricians' expert opinion

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients aged 65 or older with a history in the previous year of recurrent falls, or of a fall associated with a balance, gait, or muscle strength problem referred to the Montpellier falls prevention clinic over a 11-month period
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Serious falls | 1 day
  Falls with serious injuries are those that cause fractures, head injuries requiring admission to hospital, joint dislocations, sprains accompanied by reduced physical function, other non-specified serious joint injuries, and lacerations requiring sutures.Falls with moderate injuries are those that result in bruising, sprains, cuts, abrasions, or reduction in physical function for at least three days or in medical hel

SECONDARY OUTCOMES:
Number of Participants with injurious falls | 1 day
  A fall is defined as an "unexpected event in which the participant comes to rest on the ground, floor, or other lower level
fear of falling: Fear of falling assessed with a questionnaire to determine the number of patients not concerned, a little concerned, quite concerned or very concerned with a fear of falling | 1 day
  Fear of falling assessed with a questionnaire to determine the number of patients not concerned, a little concerned, quite concerned or very concerned with a fear of falling
mobility :Mobility assessed using a questionnaire | 1 day
  Mobility assessed using a questionnaire to determine the number of patients who, for both outside and inside displacements, do not walk, walk with a wheelchair, walk with a walker, walk with a stick, walk with a human help, or walk independently
ADLs | 1 day
  ADLs
satisfaction with the programme using a questionnaire | 1 day
  Satisfaction with the programme using a questionnaire to determine the number of patients very satisfied, somewhat satisfied, somewhat dissatisfied, or very satisfied for 6 parameters including the quality of the information provided, the suitability of recommendations, the duration of the visit, the competence of the team, and the welcoming conditions

CONTACTS AND LOCATIONS:
Overall Officials: hubert Blain, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC